CLINICAL TRIAL: NCT00000490
Title: Program on Surgical Control of Hyperlipidemias (POSCH)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: 9; R01HL049522 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Infarction; Myocardial Ischemia
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Infarction; Myocardial Ischemia | interventions — Jejunoileal Bypass; Diet, Fat-Restricted

INTERVENTIONS:
Procedure: jejunoileal bypass
Behavioral: diet, fat-restricted

SUMMARY:
To determine whether a profound reduction in serum cholesterol level, induced and maintained by partial ileal bypass, would prevent a second heart attack among men and women who had one myocardial infarction and whose blood cholesterol could not be reduced sufficiently by diet.

DETAILED DESCRIPTION:
BACKGROUND:

The correlative evidence linking elevated cholesterol to increased risk of cardiovascular disease is incontrovertible. Animal studies have shown that significant reductions in disease in humans may be forthcoming if blood lipids are reduced from elevated levels. Beginning in the 1960s, some patients had undergone a surgical bypass procedure for hyperlipidemia. Patients were selected for surgery after dietary management had been carried out for three years. The average serum cholesterol concentrations decreased markedly and the decrease was sustained.

This grant-supported clinical trial attempted to determine the effect on cardiovascular morbidity and mortality of the partial ileal bypass in patients who had suffered a myocardial infarction within the previous 5 years and who had serum cholesterol over 220 mg deciliter (200 mg if LDL cholesterol was over l40 mg).

DESIGN NARRATIVE:

Randomized, non-blind, fixed sample study with a control group and an experimental group of equal size. The experimental group received a partial ileal bypass and diet therapy to reduce serum cholesterol and triglycerides. The control group was given conventional medical therapy exclusive of cholesterol-lowering drugs. The primary endpoint was death due to any cause. Secondary endpoints included death due to atherosclerosis and morbidity from recurrent myocardial infarction, unstable angina, cerebrovascular accident. Other secondary endpoints included coronary artery bypass surgery, percutaneous transluminal coronary angioplasty, cardiac transplantation, and peripheral vascular surgery.

Beginning in January 1993, long-term morbidity and mortality follow-up are continuing through December 1997 under grant support (R01HL49522). Follow-up includes tracking morbidity and mortality by an annual telephone survey and review of patient records, including death and autopsy results. In addition, mortality and morbidity will be correlated with lipid changes and existing arteriographic results. The long-term course of control patients treated with the AHA Phase II Diet counseling will be assessed and the long-term side effects of partial ileal bypass will be evaluated.

ELIGIBILITY:
Men and women, ages 30 to 64. Had one myocardial infarction. Had hyperlipoproteinemia.

Ages: 30 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1973-06; Study Completion 1997-12

CONTACTS AND LOCATIONS:
Overall Officials: Henry Buchwald — University of Minnesota

REFERENCES:
- [Background] Buchwald H, Bourdages HR, Campos CT, Nguyen P, Williams SE, Boen JR. Impact of cholesterol reduction on peripheral arterial disease in the Program on the Surgical Control of the Hyperlipidemias (POSCH). Surgery. 1996 Oct;120(4):672-9. doi: 10.1016/s0039-6060(96)80016-x. PMID 8862377
- [Background] Buchwald H, Campos CT, Boen JR, Nguyen P, Williams SE, Lau J, Chalmers TC. Gender-based mortality follow-up from the Program on the Surgical Control of the Hyperlipidemias (POSCH) and meta-analysis of lipid intervention trials. Women in POSCH and other lipid trials. Ann Surg. 1996 Oct;224(4):486-98; discussion 498-500. doi: 10.1097/00000658-199610000-00007. PMID 8857853
- [Background] Long, JM, Brashear JR: Database Management for Clinical Trials. AFIPS Conference Proceedings: l977 National Computer Conference. AFIPS Press, Montvale, New Jersey, l977, 59-62.
- [Background] Buchwald H, Moore RB, Varco RL. Maximum lipid reduction by partial ileal bypass: a test of the lipid-atherosclerosis hypothesis. Lipids. 1977 Jan;12(1):53-8. doi: 10.1007/BF02532972. PMID 834123
- [Background] Long, JM, Brashear JR: Experience Using Standard Software to Provide a Comprehensive Information Processing System for a Large and Complex Clinical Study. Proceedings of the Second Annual Symposium on Computer Application in Medical Care. IEEE, New York, New York, l978, 563-565.
- [Background] Jelovsek FR, Bolinger RE, Davis RE, et al: Guidelines for User Access to Computerized Medical Records. J Med Systems, 2:24l-248, l978.
- [Background] Matts JP, McHugh RB. Analysis of accrual randomized clinical trials with balanced groups in strata. J Chronic Dis. 1978;31(12):725-40. doi: 10.1016/0021-9681(78)90057-7. No abstract available. PMID 748369
- [Background] Moore RB, Long JM, Matts JP, Amplatz K, Varco RL, Buchwald H. Plasma lipoproteins and coronary arteriography in subjects in the program on the surgical control of the hyperlipidemias. Preliminary report. Atherosclerosis. 1979 Feb;32(2):101-19. doi: 10.1016/0021-9150(79)90076-5. PMID 222301
- [Background] Moore RB, Buchwald H, Varco RL. The effect of partial ileal bypass on plasma lipoproteins. Circulation. 1980 Sep;62(3):469-76. doi: 10.1161/01.cir.62.3.469. PMID 7398005
- [Background] Long JM, Brashear JR, Matts JP, Bearman JE. The POSCH Information Management System: experience with alternative approaches. J Med Syst. 1980;4(3-4):355-66. doi: 10.1007/BF02222845. PMID 7264481
- [Background] Buchwald H, Moore RB, Matts JP, Long JM, Varco RL, Campbell GS, Pearce MB, Yellin AE, Blankenhorn DH, Holmes WL, Smink RD Jr, Sawin HS Jr. The Program on the Surgical Control of the Hyperlipidemias: a status report. Surgery. 1982 Oct;92(4):654-62. PMID 6750834
- [Background] Buchwald H, Rucker RD Jr., Moore RB, et al: Regression of Atherosclerosis by Surgical Cholesterol Reduction. In Noseda G et al (Eds): Lipoproteins and Coronary Atherosclerosis. Elsevier Biomedical Press, 417, 1982.
- [Background] Buchwald H, Moore RB, Varco, RL: Surgery in the Therapy of Atherosclerosis: Partial Ileal Bypass. In Atherosclerosis: Clinical Evaluation and Therapy. MTP Press Limited, International Medical Publication, 1982.
- [Background] Long JM, Brashear JR, Matts JP, et al: The Evolution of a Large Clinical Database. Proceedings of Medcomp, 82:224-229, 1982.
- [Background] Buchwald H, Fitch L, Moore RB. Overview of randomized clinical trials of lipid intervention for atherosclerotic cardiovascular disease. Control Clin Trials. 1982 Sep;3(3):271-83. doi: 10.1016/0197-2456(82)90011-3. PMID 6759035
- [Background] Buchwald H, Moore RB, Rucker RD Jr, Amplatz K, Castaneda WR, Francoz RA, Pasternak RC, Varco RL. Clinical angiographic regression of atherosclerosis after partial ileal bypass. Atherosclerosis. 1983 Jan;46(1):117-28. doi: 10.1016/0021-9150(83)90170-3. PMID 6838688
- [Background] Karnegis JN, Matts J, Tuna N, Amplatz K, Moore RB, Buchwald H. Directional ST-segment deviation in graded exercise tests correlated with motion of the individual segments of the left ventricular wall. Am J Cardiol. 1983 Sep 1;52(5):449-52. doi: 10.1016/0002-9149(83)90005-x. PMID 6613866
- [Background] Buchwald H: Intestinal Bypass for Hypercholesterolemia. In Nyhus LM (Ed.). Mastery of Surgery. Little Brown and Co., Vol II, 901-907, 1984.
- [Background] Buchwald H: Partial Ileal Bypass: A Surgical Approach to Cholesterol Lowering. In Perspectives in Lipid Disorders. McGraw-Hill Pub. Co., New York, Vol. 3, 1985.
- [Background] Buchwald H, Fitch L, Varco RL. Ileal bypass for hyperlipidemia. World J Surg. 1985 Dec;9(6):850-9. doi: 10.1007/BF01655389. No abstract available. PMID 4082609
- [Background] Karnegis JN, Matts J, Tuna N. Development and evolution of electrocardiographic Minnesota Q-QS codes in patients with acute myocardial infarction. Am Heart J. 1985 Aug;110(2):452-9. doi: 10.1016/0002-8703(85)90169-3. PMID 4025120
- [Background] Karnegis JN, Matts J, Tuna N, Amplatz K, Moore RB, Buchwald H. Quantitative assessment of left ventricular function after myocardial infarction using the minnesota Q-QS codes for resting electrocardiograms. Cathet Cardiovasc Diagn. 1985;11(4):393-400. doi: 10.1002/ccd.1810110407. PMID 3899372
- [Background] Long JM: The POSCH Secondary Intervention Trial. Proc Int Cong Prev Cardiology, Moscow, 1985.
- [Background] Long JM: Discovery and Confirmation of Causal Relationships in a Large Medical Record Database: A POSCH Experiment. Society for Clinical Trials, Annual Conference, 1985.
- [Background] Buchwald H, Fitch L, Varco RL. Surgical intervention in atherosclerosis: partial ileal bypass and the Program on Surgical Control of the Hyperlipidemias (POSCH). Pharmacol Ther. 1985;29(1):93-109. doi: 10.1016/0163-7258(85)90018-x. No abstract available. PMID 3914647
- [Background] Buchwald H, Fitch L, Varco RL: Partial Ileal Bypass; Hypercholesterolemia; Atherosclerosis. In Nyhus LM, Nelson RL (Eds.): Blackwell Scientific Publ Inc, Boston, MA, 1985, in press.
- [Background] Karnegis JN, Matts J, Tuna N, Amplatz K. Relation between Q-QS changes on the rest electrocardiogram and left ventricular function with healed myocardial infarction. Am J Cardiol. 1986 Sep 1;58(6):399-405. doi: 10.1016/0002-9149(86)90003-2. PMID 3751907
- [Background] Long JM. The POSCH data processing experience. The problem of metadata. J Med Syst. 1986 Apr;10(2):173-83. doi: 10.1007/BF00993123. PMID 3528373
- [Background] Karnegis JN, Matts J, Tuna N, Amplatz K. Comparison of exercise-positive with recovery-positive treadmill graded exercise tests. Am J Cardiol. 1987 Sep 1;60(7):544-7. doi: 10.1016/0002-9149(87)90302-x. PMID 3307368
- [Background] Buchwald H, Matts JP, Hansen BJ, Long JM, Fitch LL. Program on Surgical Control of the Hyperlipidemias (POSCH): recruitment experience. Control Clin Trials. 1987 Dec;8(4 Suppl):94S-104S. doi: 10.1016/0197-2456(87)90012-2. PMID 3440393
- [Background] Bissett JK, Matts J, Sharma B. Residual myocardial jeopardy in patients with Q-wave and non-Q-wave infarctions. Br Heart J. 1987 Nov;58(5):460-4. doi: 10.1136/hrt.58.5.460. PMID 2890362
- [Background] Campos CT, Matts JP, Fitch LL, Speech JC, Long JM, Buchwald H. Lipoprotein modification achieved by partial ileal bypass: five-year results of The Program on the Surgical Control of the Hyperlipidemias. Surgery. 1987 Aug;102(2):424-32. PMID 3303402
- [Background] Buchwald H, Campos CT. Partial ileal bypass in the therapy of familial hypercholesterolemia. Beitr Infusionsther. 1988;23:47-60. No abstract available. PMID 2461778
- [Background] Campos CT, Matts JP, Santilli SM, Fitch LL, Long JM, Speech JC, Buchwald H. Predictors of total and low-density lipoprotein cholesterol change after partial ileal bypass. Am J Surg. 1988 Jan;155(1):138-46. doi: 10.1016/s0002-9610(88)80271-x. PMID 3341527
- [Background] Campos CT, Matts JP, Fitch LL, Speech JC, Long JM, Buchwald H. Normalization of lipoproteins following partial ileal bypass in individual WHO lipoprotein phenotypes. Curr Surg. 1988 Sep-Oct;45(5):380-2. No abstract available. PMID 3073042
- [Background] Buchwald H, Matts JP, Fitch LL, Varco RL, Campbell GS, Pearce M, Yellin A, Smink RD Jr, Sawin HS Jr, Campos CT, et al. Program on the Surgical Control of the Hyperlipidemias (POSCH): design and methodology. POSCH Group. J Clin Epidemiol. 1989;42(12):1111-27. doi: 10.1016/0895-4356(89)90109-1. PMID 2685177
- [Background] Irani EA, Matts JP, Long JM, Slagle JR, and the POSCH Group: Using Artificial Neural Nets for Statistical Discovery: Observations After Using Back-Propagation, Expert Systems, and Multiple Linear Regression on Clinical Trial Data. Complex Systems, 3:295-311, 1989.
- [Background] Campos CT, Matts JP, Fitch LL, et al: Modification of Plasma Lipoproteins Following Partial Ileal Bypass. Five-Year Results of the Program of the Surgical Control of the Hyperlipidemias. In: Atherosclerosis VIII, Proceedings of the 8th International Symposium on Atherosclerosis, Rome, 9-13, October 1988; G. Crepaldi et al, (Eds), Elsevier Science Publishers B.V., Amsterdam, pp 769-774, 1989.
- [Background] Karnegis JN, Matts JP, Tuna N, Amplatz K. Estimation of left ventricular ejection fraction with healed myocardial infarction by multiple regression analysis of electrocardiographic Minnesota Q-QS codes. POSCH Group. J Electrocardiol. 1990 Jan;23(1):1-7. doi: 10.1016/0022-0736(90)90144-q. PMID 2406359
- [Background] Buchwald H, Campos CT: Partial Ileal Bypass for Control of Hyperlipidemia and Atherosclerosis. Chapter in: Gibbon's Surgery of the Chest, Fifth Edition; Sabiston DC Jr., Spencer FC (Eds); W.B. Saunders Company, Philadelphia, PA, pp 1799-1820, 1990.
- [Background] Buchwald H, Campos CT, and the POSCH Group: Preliminary Results of the Program on the Surgical Control of the Hyperlipidemias (POSCH). Chapter in: Proceedings of the 7th International Atherosclerosis and Cardiovascular Disease Meeting. Dordrecht: Kluwer Academic Publishers, in press, 1990.
- [Background] Buchwald H, Varco RL, Matts JP, Long JM, Fitch LL, Campbell GS, Pearce MB, Yellin AE, Edmiston WA, Smink RD Jr, et al. Effect of partial ileal bypass surgery on mortality and morbidity from coronary heart disease in patients with hypercholesterolemia. Report of the Program on the Surgical Control of the Hyperlipidemias (POSCH). N Engl J Med. 1990 Oct 4;323(14):946-55. doi: 10.1056/NEJM199010043231404. PMID 2205799
- [Background] Bissett JK, Ngo WL, Wyeth RP, Matts JP. Angiographic progression to total coronary occlusion in hyperlipidemic patients after acute myocardial infarction. POSCH Group. Am J Cardiol. 1990 Dec 1;66(19):1293-7. doi: 10.1016/0002-9149(90)91156-z. PMID 2244557
- [Background] Campos CT, Matts JP, Fitch LL, Speech JC, Long JM, Buchwald H. Lipid results of partial ileal bypass in patients with heterozygous, type II-A hyperlipoproteinemia. Program on the Surgical Control of the Hyperlipidemias. Surgery. 1990 Oct;108(4):601-10; discussion 610-1. PMID 2120785
- [Background] Karnegis JN, Matts JP, Tuna N, Amplatz K. Positive and negative exercise test results with and without exercise-induced angina in patients with one healed myocardial infarction: analysis of baseline variables and long-term prognosis. Am Heart J. 1991 Sep;122(3 Pt 1):701-8. doi: 10.1016/0002-8703(91)90514-i. PMID 1877445
- [Background] Obialo CI, Clayman RV, Matts JP, Fitch LL, Buchwald H, Gillis M, Hruska KA. Pathogenesis of nephrolithiasis post-partial ileal bypass surgery: case-control study. The POSCH Group. Kidney Int. 1991 Jun;39(6):1249-54. doi: 10.1038/ki.1991.158. PMID 1895677
- [Background] Matts JP, Buchwald H, Fitch LL, Campos CT, Varco RL, Campbell GS, Pearce MB, Yellin AE, Edmiston WA, Smink RD Jr, et al. Program on the Surgical Control of the Hyperlipidemias (POSCH): patient entry characteristics. The POSCH Group. Control Clin Trials. 1991 Apr;12(2):314-39. doi: 10.1016/0197-2456(91)90028-k. PMID 1645643
- [Background] Long JM, Slagle JR. Expert systems, clinical data analyses, and knowledge discovery: the POSCH AI project. Ann N Y Acad Sci. 1992 Dec 17;670:146-54. doi: 10.1111/j.1749-6632.1992.tb26085.x. No abstract available. PMID 1309084
- [Background] Karnegis JN, Matts JP, Tuna N, Hunter D, Amplatz K. Correlation of coronary with peripheral arterial stenosis. The POSCH Group. Atherosclerosis. 1992 Jan;92(1):25-30. doi: 10.1016/0021-9150(92)90006-3. PMID 1575819
- [Background] Buchwald H, Campos CT, Matts JP, Fitch LL, Long JM, Varco RL. Women in the POSCH trial. Effects of aggressive cholesterol modification in women with coronary heart disease. The POSCH Group. Program on the Surgical Control of the Hyperlipidemias. Ann Surg. 1992 Oct;216(4):389-98; discussion 398-400. doi: 10.1097/00000658-199210000-00001. PMID 1417188
- [Background] Buchwald H, Matts JP, Fitch LL, Campos CT, Sanmarco ME, Amplatz K, Castaneda-Zuniga WR, Hunter DW, Pearce MB, Bissett JK, et al. Changes in sequential coronary arteriograms and subsequent coronary events. Surgical Control of the Hyperlipidemias (POSCH) Group. JAMA. 1992 Sep 16;268(11):1429-33. PMID 1512911
- [Background] Buchwald H, Fitch LL, Matts JP, Johnson JW, Hansen BJ, Stuenkel MR, Brooks HB. Perception of quality of life before and after disclosure of trial results: a report from the Program on the Surgical Control of the Hyperlipidemias (POSCH). Control Clin Trials. 1993 Dec;14(6):500-10. doi: 10.1016/0197-2456(93)90030-h. PMID 8119065
- [Background] Matts JP, Karnegis JN, Campos CT, Fitch LL, Johnson JW, Buchwald H. Serum creatinine as an independent predictor of coronary heart disease mortality in normotensive survivors of myocardial infarction. POSCH Group. J Fam Pract. 1993 May;36(5):497-503. PMID 8482933
- [Background] Bissett JK, Wyeth RP, Matts JP, Johnson JW. Plasma lipid concentrations and subsequent coronary occlusion after a first myocardial infarction. The POSCH Group. Am J Med Sci. 1993 Mar;305(3):139-44. doi: 10.1097/00000441-199303000-00002. PMID 8447332
- [Background] Fitch LL, Buchwald H, Matts JP, Johnson JW, Campos CT, Long JM. Effect of aspirin use on death and recurrent myocardial infarction in current and former cigarette smokers. Program on the Surgical Control of the Hyperlipidemias Group. Am Heart J. 1995 Apr;129(4):656-62. doi: 10.1016/0002-8703(95)90311-9. PMID 7900613
- [Background] Buchwald H, Campos CT. Control of risk factors in atherosclerosis. POSCH Report. Ann N Y Acad Sci. 1995 Jan 17;748:342-55; discussion 355-6. doi: 10.1111/j.1749-6632.1994.tb17331.x. No abstract available. PMID 7695177
- [Background] Matts JP, Buchwald H, Fitch LL, Campos CT, Varco RL, Campbell GS, Pearce MB, Yellin AE, Smink RD Jr, Sawin HS Jr, et al. Subgroup analyses of the major clinical endpoints in the Program on the Surgical Control of the Hyperlipidemias (POSCH): overall mortality, atherosclerotic coronary heart disease (ACHD) mortality, and ACHD mortality or myocardial infarction. J Clin Epidemiol. 1995 Mar;48(3):389-405. doi: 10.1016/0895-4356(94)00145-g. PMID 7897460
- [Background] Campos CT, Buchwald H, and the POSCH Group: The Program on the Surgical Control of the Hyperlipidemias (POSCH): Demonstration of the Beneficial Effects of Treatment of Hypercholesterolemia. Cardiovasc Risk Factors, 2:261-275, 1992.
- [Background] Buchwald H, Campos CT, Boen JR, Nguyen PA, Williams SE. Disease-free intervals after partial ileal bypass in patients with coronary heart disease and hypercholesterolemia: report from the Program on the Surgical Control of the Hyperlipidemias (POSCH). J Am Coll Cardiol. 1995 Aug;26(2):351-7. doi: 10.1016/0735-1097(95)80006-3. PMID 7608434
- [Background] Buchwald H, Varco RL, Boen JR, Williams SE, Hansen BJ, Campos CT, Campbell GS, Pearce MB, Yellin AE, Edmiston WA, Smink RD Jr, Sawin HS Jr. Effective lipid modification by partial ileal bypass reduced long-term coronary heart disease mortality and morbidity: five-year posttrial follow-up report from the POSCH. Program on the Surgical Control of the Hyperlipidemias. Arch Intern Med. 1998 Jun 8;158(11):1253-61. doi: 10.1001/archinte.158.11.1253. PMID 9625405
- [Background] Gould AL, Cariski AT. Meta-analysis by the Program on the Surgical Control of the Hyperlipidemias (POSCH) investigators. Ann Surg. 1998 Feb;227(2):314-6. doi: 10.1097/00000658-199802000-00031. No abstract available. PMID 9488536
- [Background] Buchwald H, Hunter DW, Tuna N, Williams SE, Boen JR, Hansen BJ, Titus JL, Campos CT. Myocardial infarction and percent arteriographic stenosis of culprit lesion: report from the Program on the Surgical Control of the Hyperlipidemias (POSCH). Atherosclerosis. 1998 Jun;138(2):391-401. doi: 10.1016/s0021-9150(98)00049-5. PMID 9690924
- [Background] Buchwald H, Boen JR, Nguyen PA, Williams SE, Matts JP. Plasma lipids and cardiovascular risk: a POSCH report. Program on the Surgical Control of the Hyperlipidemias. Atherosclerosis. 2001 Jan;154(1):221-7. doi: 10.1016/s0021-9150(00)00467-6. PMID 11137103